CLINICAL TRIAL: NCT04048226
Title: The Effect of Intraoperative Dexmedetomidine-Ketamine Infusion on the Patients Undergoing Radical Mastectomy: Randomized Controlled Study
Brief Title: Dexmedetomidine-Ketamine Infusion in Breast Surgeries
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Dr, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 33108/05/19; Tanta University (Other: Faculty of Medicine, Tanta University)
Record Dates: First submitted 2019-08-06; First posted 2019-08-07 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Total Intravenous Anesthesia
Keywords: Dexmedetomidine; Ketamine; Radical Mastectomy; Chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Anesthesia, Intravenous

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: * The patients will be blind through the use of closed sealed envelops.
  * The investigator will be blind through the use of syringe pump containing normal saline in the control group by the aid of anesthesia resident who will not participate in the study.
  * The measurement will be collected by anesthesia nurse not participating in the study and blinded to its group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): The patients in this group will be connected to the syringe pump that contain normal saline with starting infusion at a rate of 0.1 ml/kg/hr till the end of the surgery.
  Interventions: Drug: Placebos
- Dexmedetomidine-Ketamine group (Experimental): The patients in this group will be connected to the syringe pump that contain mixture of dexmedetomidine and ketamine with starting infusion at a rate of 0.1 ml/kg/hr till the end of the surgery. The solution will contain 2 ug dexmedetomidine/ml and 1 mg ketamine/ml.
  Interventions: Drug: Dexmedetomidine +Ketamine

INTERVENTIONS:
Drug: Placebos — The patients in this group will be connected to the syringe pump that contain normal saline with starting infusion at a rate of 0.1 ml/kg/hr till the end of the surgery.
  Other Names: Normal saline infusion
  Arms: Control group
Drug: Dexmedetomidine +Ketamine — The patients in this group will be connected to the syringe pump that contain mixture of dexmedetomidine and ketamine with starting infusion at a rate of 0.1 ml/kg/hr till the end of the surgery. The solution will contain 2 ug dexmedetomidine/ml and 1 mg ketamine/ml.
  Other Names: Intravenous anesthesia
  Arms: Dexmedetomidine-Ketamine group

SUMMARY:
* This is a prospective randomized double blind controlled study.
* Female patients undergoing radical mastectomy will be included in this study where they will be randomly allocated into; - Control group in which patients will receive continuous infusion of normal saline.

Dexmedetomidine-Ketamine group in which patients will receive continuous infusion of ketamine and dexmedetomidine.

The intraoperative and postoperative opioid consumption will be measured. Also, the postoperative pain score and the incidence of chronic pain will be assessed.

DETAILED DESCRIPTION:
This prospective randomized controlled study will be carried out on 70 female patients who will be presented for radical mastectomy in the general surgery department in Tanta university hospitals over three month duration and 6 months follow up that starts immediately after obtaining ethical committee approval, an informed written consent will be obtained from all the participants, all patients data will be confidential and will be used for the current study only.

-Inclusion criteria: Female patients aged 50-70 years, ASA class I-III, and presented for elective radical mastectomy.

- Exclusion criteria: Patients refused to participate. Patients with known or suspected or known allergy to the used medication. Patients with preoperative chronic pain, Patients received preoperative opioids or gabapentoids. Patients with major cardiac, renal, respiratory, or hepatic disease. Uncooperative patients. Obese patients with BMI >36

Anesthetic technique Once the patients will arrive to the operating room, intravascular access will be established, fluid preload will be started, and basic monitor will be attached. An assistant anesthetist will help in preparation of a 50 ml syringe connected to a syringe pump that will contain normal saline or a mixture of 100 ug dexmedetomidine and 50 mg ketamine.

Anesthesia will be induced by fentanyl 1 ug/kg, propofol 1.5 mg/kg, and cis-atracurium 0.15 mg/kg to facilitate tracheal intubation. After endotracheal intubation, the patients will be connected to a mechanical ventilator with its parameters adjusted to maintain etCo2 32-36 mmHg. Anesthesia will be maintained by isoflurane 1% MAC in mixture of oxygen:air 1:1 with the use of low flow (1 ml/min). The patients will be randomly allocated into two equal groups by the aid of computer-generated software of randomization: -

• Control group (35 patients): The patients in this group will be connected to the syringe pump that contain normal saline with starting infusion at a rate of 0.1 ml/kg/hr till the end of the surgery.

• Dexmedetomidine-Ketamine group (35 patients): The patients in this group will be connected to the syringe pump that contain mixture of dexmedetomidine and ketamine with starting infusion at a rate of 0.1 ml/kg/hr till the end of the surgery. The solution will contain 2 ug dexmedetomidine/ml and 1 mg ketamine/ml.

All the patients will be connected to a bispectral index monitor with maintaining its value ranging 40-60. Increase in the BIS value over 60 will be managed by additional dose of fentanyl 0.5 ug/kg till decrease the BIS below 60. If the BIS is still over 60, increasing the isoflurane 0.2 % MAC till it decreased below 60.

At the end of the surgery, switching off the inhalational anesthetics, reversal of muscle relaxation, and awake tracheal extubation will be done with transporting the patients to the PACU for postoperative follow up and monitoring.

- Measurements:

1. Patient age, weight, height.
2. Morphine consumption in the first 24 h postoperatively.
3. The total dose consumption of fentanyl consumed intraoperatively.
4. The total volume consumed of isoflurane intraoperatively (ml/hr).
5. The postoperative Visual Analogue Score (VAS): It will be measured every 2 hours till 8 h, then every 4 h till 24 h. In case of increase the VAS more than 3, a rescue analgesia will be administrated in the form of 3 mg morphine i.v that may be repeated.
6. The time for the first request of morphine rescue analgesia
7. The incidence of chronic pain (Follow up of the patients will be carried out in the pain clinic after discharge from hospital every 2 weeks for a period of 6 months for assessment of the incidence of postoperative chronic pain.
8. The recovery profile
9. The incidence of complications

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 50-70 years, ASA class I-III, and presented for elective radical mastectomy.

Exclusion Criteria:

* Patients refused to participate.
* Patients with known or suspected or known allergy to the used medication.
* Patients with preoperative chronic pain,
* Patients received preoperative opioids or gabapentoids.
* Patients with major cardiac, renal, respiratory, or hepatic disease.
* Uncooperative patients.
* Obese patients with BMI >36

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is not based on self-representation of gender identity.
Enrollment: 103 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2024-03-20 (Actual)

PRIMARY OUTCOMES:
The postoperative morphine consumption | The first 24 hours postoperatively
  The total dose of morphine consumed postoperative as a rescue analgesia to maintain the VAS less than 4

SECONDARY OUTCOMES:
The intraoperative fentanyl consumption | Through out the whole intraoperative period
  The intraoperative consumption of fentanyl
Incidence of the chronic pain | 6 months after the surgery
  The patients who suffer from chronic pain during 6 months of follow up using simple questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Principal Investigator — Lecturer of Anesthesia and Intensive Care, Tanta University
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers.